CLINICAL TRIAL: NCT01707797
Title: Predicting Caries Risk in Underserved Toddlers in Primary Healthcare Settings A Stratified (by Race, Ethnicity, and Medicaid Status) Study to Develop a Caries Risk Prediction Questionnaire
Brief Title: Predicting Caries Risk in Underserved Toddlers in Primary Healthcare Settings
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Margherita Fontana, DDS, PhD, Professor Cariology Discipline Co-coordinator, University of Michigan
Other Study IDs: NIDCR 11-101; U01DE021412-01A1 (NIH)
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Dental Caries
Keywords: dental caries; high risk; dental cavities; children dental care
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy children aged 9-15 months: Healthy children aged 12 months (± 3 months) at baseline stratified by Medicaid status and/or race/ethnicity to ensure a diverse representation. Each child will be paired with the primary caregiver, whom the investigators expect to most likely be the adult parent or legal guardian.

SUMMARY:
The study aims to develop a questionnaire that can be used to help uncover a child's risk of developing dental caries (also known as tooth decay or a cavity). The aim is to develop a practical and easily-scored risk tool that a primary medical care provider can use to help find young children with the highest risk for developing cavities.

DETAILED DESCRIPTION:
The duration of expected time to participate is 3 years (which includes 3 dental examinations).

ELIGIBILITY:
Inclusion Criteria:

Adults

* If Primary Caregiver is the Parent/Legal guardian: The parent/legal guardian must provide written informed consent for the child and her/himself (if s/he is the primary caregiver) prior to participation.
* If Primary Caregiver is not the Parent/Legal Guardian: If another individual is the primary caregiver, then this individual must provide written informed consent for her/himself prior to participation.
* The parent/legal guardian and the participating primary caregiver must each be at least 18 years old or an emancipated minor
* The parent/legal guardian must consent and allow examination of the oral cavity of her/his child. The primary caregiver must complete the caries risk assessment questionnaire.
* The primary caregiver must be willing to participate, anticipate being the child's primary caregiver during the study period, and anticipate being available for all examinations (baseline, 18 month follow up, and 36 month follow up), in addition to intermediate contacts in between examinations.

Children

* Child must be 9-15 months of age at the time of the baseline study visit.
* Child must be generally healthy (i.e., no current medical condition that makes it difficult for her/him to receive a dental examination).
* Child must allow examination of the oral cavity.

Exclusion Criteria:

Adults

* A participant pair (adult-child) who demonstrates an inability to comply with study protocol requirements will be excluded - this determination will be at the Site Primary Investigator's discretion.
* Non-English, non-Spanish reading/speaking individuals will be excluded, as they will not be able to comprehend the consent document or complete the risk questionnaire.

Children

* Children who are in foster care at study initiation will be excluded, due to the likelihood that their primary caregiver will change multiple times during the length of the study.
* Need for antibiotic and/or sedative premedication prior to dental exam.
* Uncontrolled epilepsy.
* Active cancer treatment.
* Unrepaired congenital heart defects that would require premedication prior to dental exam.

Ages: 9 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged 12 months (± 3 months) at baseline stratified by Medicaid status and/or race/ethnicity to ensure a diverse representation. Each child will be paired with the primary caregiver, whom the investigators expect to most likely be the adult parent or legal guardian.
Sampling Method: Probability Sample
Enrollment: 1326 (Actual)
Dates: Start 2012-11-15 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Presence of any caries at baseline and incidence and/or progression of any caries lesions at follow up examinations | 3 years
  Outcomes will be defined at the participant level.
  1. Presence of any caries at baseline (defined as ICDAS ≥ 3, filling, or missing due to caries).
  2. Incidence (ICDAS ≥ 3, filling, or missing due to caries) and/or progression (change from ICDAS= 3 or 4 to ICDAS=5 or 6, or filling, or missing due to caries) of any caries lesions at the follow-up examinations.

SECONDARY OUTCOMES:
Presence of any caries at baseline | Baseline
  Presence of any caries at baseline (defined as ICDAS > 0, which includes all early caries, filling, or missing due to caries). Presence of any caries at baseline (defined as ICDAS ≥ 5, which includes only frank cavitation, filling, or missing due to caries)
Incidence and/or progression of any caries lesions at the follow-up examinations. | 3 years
  Incidence and/or progression of any caries lesions at the follow-up examinations. Progression is defined as change from ICDAS=0 to ICDAS=1 or higher, or filling, or missing due to caries; change from ICDAS=1 or 2 to ICDAS=3 or higher, or filling, or missing due to caries; or change from ICDAS=3 or 4 to ICDAS=5 or 6, or filling, or missing due to caries.
  Incidence of any caries lesions at the follow-up examinations. Because only distinct cavitation is included at baseline, no progression outcomes from baseline to follow-up will be defined.
counts of the number of carious surfaces | 3 years
  1. Counts of the number of carious surfaces (dmfs), using ICDAS ≥ 3 to define decayed surfaces.
  2. Counts of the number of carious surfaces (dmfs), using ICDAS > 0 to define decayed surfaces.
  3. Counts of the number of carious surfaces (dmfs), using ICDAS ≥ 5 to define decayed surfaces

CONTACTS AND LOCATIONS:
Overall Officials: Margherita Fontana, DDS, PhD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Indiana University Oral Health Research Institute, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Duke Health Center, Durham, North Carolina

REFERENCES:
- [Derived] Fontana M, Eckert GJ, Keels MA, Jackson R, Katz BP, Kemper AR, Levy BT, Levy SM, Yanca E, Kelly S, Daly JM, Patterson B, McKnight P. Predicting Caries in Medical Settings: Risk Factors in Diverse Infant Groups. J Dent Res. 2019 Jan;98(1):68-76. doi: 10.1177/0022034518799080. Epub 2018 Sep 11. PMID 30205016
- [Derived] Fontana M, Eckert GJ, Keels MA, Jackson R, Katz B, Levy BT, Levy SM. Fluoride Use in Health Care Settings: Association with Children's Caries Risk. Adv Dent Res. 2018 Feb;29(1):24-34. doi: 10.1177/0022034517735297. PMID 29355412